CLINICAL TRIAL: NCT03498846
Title: Modified Corneal Epithelial Autograft With Middle Lamellar Keratoplasty for Severe Corneal Burn
Brief Title: Modified Corneal EA With Middle LKP for Severe Corneal Burn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Clinical investigator, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018KYPJ070
Record Dates: First submitted 2018-04-07; First posted 2018-04-17 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Corneal Burn
MeSH Terms: conditions — Eye Burns

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified EA and AMLK (Experimental): Modified corneal epithelial autograft (EA) combined with allogeneic middle lamellar keratoplasty (AMLK) is used for the treatment of patients with severe corneal burn.
  Interventions: Procedure: Modified EA and AMLK
- LA and AMLK (Active Comparator): Limbal autograft (LA) combined with AMLK is used for the treatment of patients with severe corneal burn.
  Interventions: Procedure: LA and AMLK

INTERVENTIONS:
Procedure: Modified EA and AMLK — Two pieces of corneal epithelial tissue with 2mmx3mm will be obtained from the fellow eye using femtosecond laser technology. This epithelial autograft (EA) is then ready for transplantation on the disease eye, following the procedure of allogeneic middle lamellar keratoplasty (AMLK).
  Arms: Modified EA and AMLK
Procedure: LA and AMLK — A 3-clock-hour limbal autograft (LA) will be obtained from the fellow eye. This is then ready for transplantation on the disease eye following the procedure of AMLK.
  Arms: LA and AMLK

SUMMARY:
The purpose of this pilot study is to explore whether modified corneal epithelial autograft (EA) combined with allogeneic middle lamellar keratoplasty (AMLK) is more effective than limbal autograft (LA) with AMLK for ocular surface reconstruction in patients with severe corneal burn.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral severe corneal burn with more than half limbal stem cells deficiency (LSCD). The history of the disease is at least 12 months at the time of screening visit.
2. Presence of superficial neo-vascularization affecting at least 2 cornea quadrants and involving central cornea.
3. Informed consent signed by a patient or legal guardian, or having the ability to comply with study assessments for the full duration of the study.

Exclusion Criteria:

1. LSCD of mild degree, with less than 2 quadrants of neo-vessel invasion and without central cornea involvement.
2. LSCD by ocular surface disorders other than ocular burns.
3. Eyelids malposition.
4. The center corneal thickness<450µm, the depth of corneal opacity<150µm or the full corneal lamellar opacity.
5. High myopia with a spherical equivalent of -15.0 D or less.
6. Corneal or ocular surface infection within 30 days prior to study entry.
7. Ocular surface malignancy.
8. Uncontrolled diabetes with most recent HgA1c greater than 8.5%.
9. Renal failure with creatinine clearance ≤ 25mL/min per 1.73 m2.
10. Alanine aminotransferase > 40IU/L, or aspartate aminotransferase > 40IU/L.
11. Platelet levels < 150,000 or > 450,000 per microliter.
12. Hemoglobin < 12.0 g/dL (male) or < 11.0 g/dL (female);
13. Prothrombin time > 16s and activated partial thrombin time > 35s in patients not accepting anticoagulant therapy; An international normalized ratio greater than 3 in patients accepting anticoagulant therapy.
14. Pregnancy (positive test) or lactation.
15. Participation in another simultaneous medical investigation or clinical trial.
16. Severe cicatricial eye disease; Conjunctival scarring with fornix shortening.
17. Ocular comorbidities that affect the prognosis of transplantation, such as advanced glaucoma or retinal diseases.
18. Severe dry eye disease as determined by Schirmer's test < 2mm at least in one eye.
19. Any medical or social condition that in the judgment of the investigator would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent.
20. Signs of current infection, including fever and treatment with antibiotics.

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-12-09 (Estimated); Study Completion 2020-05-09 (Estimated)

PRIMARY OUTCOMES:
Success rate of corneal reepithelialization in disease eyes | 12 months
  The success rate of patients with completely epithelized and avascular corneal surface in disease eyes

CONTACTS AND LOCATIONS:
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China